CLINICAL TRIAL: NCT00367744
Title: Placebo Controlled Study of Rosiglitazone in HIV Lipoatrophy
Brief Title: Rosiglitazone Effect on Mitochondria and Lipoatrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI060484-02-C; AI060484-C (Other Grant/Funding Number: NIAID)
Record Dates: First submitted 2006-08-21; First posted 2006-08-23 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2006-08

CONDITIONS: HIV Infections
Keywords: mitochondria; HIV; lipoatrophy
MeSH Terms: conditions — HIV Infections; Lipodystrophy | interventions — Rosiglitazone; Thiazolidinediones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosigitazone arm (Active Comparator): Rosiglitazone active 4 mg BID
  Interventions: Drug: Rosiglitazone
- Placebo arm (Placebo Comparator): Matching Placebo BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosiglitazone — Rosiglitazone 4mg BID
  Other Names: Glitazones, avandia
  Arms: Rosigitazone arm
Drug: Placebo — Placebo for rosiglitazone
  Arms: Placebo arm

SUMMARY:
The purpose of this study is to examine the effect of rosiglitazone on limb fat and mitochondrial indices in HIV-1-infected subjects receiving stable antiretroviral therapy that does not contain stavudine (d4T) or zidovudine (AZT).

DETAILED DESCRIPTION:
This is a phase II, randomized, double-blind, placebo-controlled study of rosiglitazone for the treatment of HIV-associated lipoatrophy. Subjects will receive blinded study treatment for 48 weeks. This study will examine the effect of rosiglitazone on limb fat and mitochondrial indices in HIV-1-infected subjects receiving stable antiretroviral therapy that does not contain d4T or AZT. The study also will assess the safety and tolerability of rosiglitazone in this population, and its effect on carotid IMT, prevalence of metabolic syndrome, lipid parameters and glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Lipoatrophy
* Thymidine sparing ARV for at least 24 weeks
* Prior thymidine NRTIs for at least 12 months

Exclusion Criteria:

* Diabetes
* Heart failure
* Liver disease
* Hormonal therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2006-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace McComsey, Principal Investigator — Case Western Reserve University
Locations (2):
- United States (2):
  - Cleveland Clinc Foundation, Cleveland, Ohio
  - University Hospitals of Cleveland/Case Western Reserve University, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tungsiripat M, El-Bejjani D, Rizk N, Dogra V, O'Riordan MA, Ross AC, Hileman C, Storer N, Harrill D, McComsey GA. Carotid intima media thickness, inflammatory markers, and endothelial activation markers in HIV Patients with lipoatrophy increased at 48 weeks regardless of use of rosiglitazone or placebo. AIDS Res Hum Retroviruses. 2011 Mar;27(3):295-302. doi: 10.1089/aid.2010.0187. Epub 2010 Oct 23. PMID 20969457
- [Derived] Tungsiripat M, Bejjani DE, Rizk N, O'riordan MA, Ross AC, Hileman C, Storer N, Harrill D, McComsey GA. Rosiglitazone improves lipoatrophy in patients receiving thymidine-sparing regimens. AIDS. 2010 Jun 1;24(9):1291-8. doi: 10.1097/QAD.0b013e328339e274. PMID 20453626
- See also: to find more about rosiglitazone effectiveness on Lipoatrophy — https://www.ncbi.nlm.nih.gov/pubmed/20453626

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited at Case Western Reserve University and Cleveland Clinic. Recruitment occurred between from July 2006 (first subject was randomized) to December 2007 (last subject was randomized).
Pre-assignment Details: A total of 71 subjects were randomized. Results are reported for 71 subjects.
Groups:
- Rosiglitazone: Rosiglitazone 4 mg daily for 4 weeks then the dose was increased to 4mg twice daily for the remainder of the study (44 weeks)
- Placebo: Placebo arm for the whole duration of the study
Period: Overall Study
Arm/Group | Rosiglitazone | Placebo
Started | 34 | 37
Completed | 30 | 32
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Rosiglitazone: Rosiglitazone 4mg daily for 4 weeks then the dose increased to 4mg twice daily for the remainder of the study (44 weeks)
- Placebo: Placebo arm
- Total: Total of all reporting groups
Arm/Group | Rosiglitazone | Placebo | Total
Number analyzed (Participants) | 34 | 37 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 37 | 71
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (7) | 50 (7) | 49.04 (7)
Gender [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 29 | 30 | 59
Region of Enrollment [Number; unit: participants]
  United States | 34 | 37 | 71
CD4+ cell count [Median (Inter-Quartile Range); unit: cells/mm3] | 596 [437 to 706] | 691 [423 to 861] | 645.5 [430 to 787]

OUTCOME MEASURES:

1. Primary Outcome: Change in Limb Fat at 48 Weeks
Description: Limb fat was measured at baseline and visit week 48 using dual-energy x-ray absorptiometry (DEXA), and change from baseline to week 48 (week 48 - baseline) was estimated for the treatment groups.
Time Frame: 48 weeks
Population: Intention to treat analysis with last observation carried forward if week 48 limb fat data was missing and post-baseline limb fat was availble.
Measure: Median (Inter-Quartile Range); unit: grams
Groups:
- Rosiglitazone: Rosiglitazone 4mg daily for 4 weeks then BID for 44 weeks
Arm/Group | Rosiglitazone | Placebo
Number analyzed (Participants) | 34 | 37
grams | 448 [138 to 1670] | 153 [-100 to 682]
Statistical Analysis 1: Comparison: Rosiglitazone vs Placebo; The primary outcome measure was the change in limb fat at 48 weeks between the rosiglitazone and placebo group; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney); Treatment groups were compared for change in limb fat using a two-sided signed rank test

2. Secondary Outcome: the Change in the Carotid IMT of the Common Carotid Artery
Description: Carotid IMT of the Common carotid artery (CCA) was measured at baseline and week 48, and change from baseline to week 48 (week 48 - baseline) was estimated for the treatment groups.
Time Frame: 48 weeks
Population: Intention to treat analysis with last observation carried forward if week 48 carotid IMT data was missing and post-baseline IMT data was available
Measure: Median (Inter-Quartile Range); unit: mm
Groups:
- Rosiglitazone: Rosiglitazone 4mg daily for 4 weeks then 4mg BID for 44 weeks
Arm/Group | Rosiglitazone | Placebo
Number analyzed (Participants) | 30 | 32
mm | 0.10 [-0.05 to 0.25] | 0.15 [0 to 0.25]

ADVERSE EVENTS:
Time Frame: weeks 2,4,12,18,24,36 and 48
Description: assessment for adverse events were done at study visits (weeks 24, and 48) additional safety visits occurred at weeks 2,4,12,18 and 36
Arm/Group | Rosiglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 15/34 | 13/37
Other Adverse Events (participants affected / at risk) | 6/34 | 7/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosiglitazone (N=34) | Placebo (N=37)
Elevated Cholesterol (Grade 2 or 3) (Cardiac disorders) | 4 | 6
Elevated Triglycerides (Grade 2) (Blood and lymphatic system disorders) | 4 | 1
Elevated LDL Cholesterol (Grade 2 or 3) (Vascular disorders) | 0 | 4
Elevated Blood Pressure (Grade 2 or 3) (Vascular disorders) | 5 | 2
Low ANC (Grade 2) (Blood and lymphatic system disorders) | 2 | 1
Low Phosphate (Grade 2 or 3) (Musculoskeletal and connective tissue disorders) | 4 | 2
Elevated Creatinine (Grade 2) (Blood and lymphatic system disorders) | 7 | 7
Irregular Pulse (Cardiac disorders) | 1 | 0
Elevated AST (Grade 2) (Hepatobiliary disorders) | 0 | 1
Elevated ALT (Hepatobiliary disorders) | 1 | 1
Angina (Cardiac disorders) | 1 | 0
Elevated Glucose (Grade 2) (Blood and lymphatic system disorders) | 1 | 0
Decreased Platelets (Grade 2 or 3) (Blood and lymphatic system disorders) | 1 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Depression (Grade 2) (Psychiatric disorders) | 0 | 1
Suicidal Gesture (Grade 4) (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosiglitazone (N=34) | Placebo (N=37)
Low Fasting Glucose (Grade 1) (Metabolism and nutrition disorders) | 1 | 0
Low Phosphate (Grade 2) (Musculoskeletal and connective tissue disorders) | 5 | 5
Elevated Bilirubin (Grade 2 or 3) (Blood and lymphatic system disorders) | 0 | 1
Elevated Creatine Kinase (Grade 2) (Musculoskeletal and connective tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Limitations of the study include a relative small sample size as well as loss of follow up of 9 participants at the end of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No